CLINICAL TRIAL: NCT03115112
Title: A Phase 3, Randomized, Double-Blind, Active-Controlled Study to Evaluate the Effects of Bexagliflozin Versus Sitagliptin in Subjects With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control by Metformin
Brief Title: Safety and Efficacy of Bexagliflozin Compared to Sitagliptin as Add-on Therapy to Metformin in Type 2 Diabetes Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Theracos (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THR-1442-C-423
Record Dates: First submitted 2017-04-11; First posted 2017-04-14 (Actual); Results first posted 2021-06-04 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — bexagliflozin; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bexagliflozin (Active Comparator): Subjects will receive a bexagliflozin tablet, 20 mg, once daily for the duration of the study. Subjects will continue taking metformin and receive placebo for sitagliptin daily for the duration of the study.
  Interventions: Drug: Bexagliflozin; Drug: Placebo for sitagliptin
- Sitagliptin (Active Comparator): Subjects will receive a sitagliptin tablet, 100 mg, once daily for the duration of the study. Subjects will continue taking metformin and receive placebo for bexagliflozin for the duration of the study.
  Interventions: Drug: Sitagliptin; Drug: Placebo for bexagliflozin

INTERVENTIONS:
Drug: Bexagliflozin — tablets containing 20 mg bexagliflozin
  Other Names: EGT0001442, EGT0001474
  Arms: Bexagliflozin
Drug: Sitagliptin — tablets containing 100 mg sitagliptin
  Other Names: Januvia
  Arms: Sitagliptin
Drug: Placebo for sitagliptin — inactive tablets to match the appearance of sitagliptin tablets
  Arms: Bexagliflozin
Drug: Placebo for bexagliflozin — inactive tablets to match the appearance of bexagliflozin tablets
  Arms: Sitagliptin

SUMMARY:
The purpose of this study is to investigate the effect of bexagliflozin compared to sitagliptin as an add-on therapy to metformin in lowering hemoglobin A1c (HbA1c) levels in subjects with type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
This was a phase 3, multi-center, randomized, double-blind, parallel-group study to demonstrate that bexagliflozin was non-inferior to sitagliptin as add-on therapy in subjects whose T2DM was not adequately controlled by metformin treatment alone. The primary effectiveness endpoint was the change in HbA1c from baseline at week 24.

At the time of screening, all subjects were to have taken metformin at a stable dose of ≥ 1500 mg per day for ≥ 8 weeks and have received diet and exercise counseling. A total of 374 eligible subjects were to be enrolled in the study. Subjects who successfully completed a 1-week run-in and who met all eligibility criteria were to be randomized in a 1:1 ratio to receive once daily double-blind treatment of either active bexagliflozin tablets with placebo sitagliptin tablets or placebo bexagliflozin tablets and active sitagliptin tablets. The study subjects were to continue receiving open-labeled metformin during the entire study at a stable dose and frequency. The treatment period was 24 weeks and was conducted in an outpatient setting.

Randomization was stratified by HbA1c (≤ 8.5% vs. ˃ 8.5%) values. Symptoms and blood sugars related to the occurrence of hyperglycemia, hypoglycemic events or symptoms that could indicate ketoacidosis were to be recorded. Bexagliflozin tablets, 20 mg or placebo, and sitagliptin tablets, 100 mg or placebo, were to be taken once daily at approximately the same time each day either before or after breakfast. Background metformin was to be taken at the same dose and frequency from screening throughout the entire study.

Each subject was advised to return to the clinic at weeks 6, 12, 18 and 24 for efficacy assessment and safety monitoring, including review of AEs and concomitant medication, vital signs, ECG, physical examination and blood and urine specimen collections. Subjects were to return to the clinic for a follow-up exit visit at week 26 or 2 weeks after the last dose of study drugs if subjects withdrew from the study prior to week 24.

ELIGIBILITY:
Each subject was required to meet the following criteria at the time of enrollment to be eligible for the study:

1. To have been male or female adults ≥ 18 years of age.
2. To have been negative on the urine pregnancy test and agreed to abstain from coitus or use contraception during the entire study if a subject was female of childbearing potential.
3. To have had a diagnosis of T2DM with HbA1c levels between 7.0% and 11% (inclusive) at the time of screening.
4. To have been treated with a stable dose of ≥ 1500 mg/day metformin only along with diet and exercise counseling for at least 8 weeks at the time of screening.
5. To have had a BMI ≤ 45 kg per m2 at the time of screening.
6. To have been taking stable doses of treatment for dyslipidemia and/or hypertension for 30 days if applicable.
7. To have been willing and able to return for all clinic visits and to complete all study-required procedures.
8. To have adhered to the investigational product administration requirements as evidenced by missing no more than 1 day of run-in medications.

Potential subjects who exhibited any of the following characteristics were to be excluded from the study:

1. Diagnosis of type 1 diabetes mellitus or maturity-onset diabetes of the young (MODY)
2. Hemoglobinopathy that affected HbA1c measurement
3. Any contraindication to the safe use of DPP-4 therapy or sitagliptin, including known hypersensitivity reaction
4. History of pancreatitis
5. Genitourinary tract infection within 6 weeks of screening or history of ≥ 3 genitourinary infections requiring treatment within 6 months from the time of screening
6. Cancer, active or in remission, for < 3 years
7. History of alcohol or illicit drug abuse in the past 2 years
8. Triglycerides > 500 mg dL-1 at Visit V1
9. Evidence of abnormal liver function tests (total bilirubin or alkaline phosphatase > 1.5 x upper limit of normal (ULN) with the exception of isolated Gilbert's syndrome); or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 x ULN
10. Estimated GFR, as calculated by the modification of diet in renal disease study equation (MDRD), < 60 mL min-1 per 1.73 m2 at the time of screening.
11. Uncontrolled hypertension (SBP > 160 mm Hg or diastolic BP > 95 mm Hg) at Visit V1
12. Life expectancy < 2 years
13. History of MI, unstable angina, stroke or hospitalization for heart failure within 3 months at the time of screening
14. History of treatment with an investigational drug within 30 days or within 7 half-lives of the investigational drug, whichever is longer
15. Previous treatment with bexagliflozin or EGT0001474 study drug
16. Currently or within 3 months of taking any SGLT2 inhibitor
17. Currently participating in another interventional trial
18. Prior renal transplantation or evidence of nephrotic syndrome (defined as a urine albumin-to-creatinine ratio (UACR) > 1500 mg g-1 at the time of screening).
19. Any condition, disease, disorder or clinically relevant abnormality that could have jeopardized the subject's appropriate participation in this study or obscure the effects of treatment
20. Female subjects who were pregnant or nursing
21. Two or more consecutive SMBG measures ≥ 250 mg dL-1 (13.9 mmol L-1) prior to randomization accompanied by clinical signs or symptoms of hyperglycemia prior to randomization, including weight loss, blurred vision, increased thirst increased urination, or fatigue

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Paul Lock, MD, Study Director — Theracos Sub, LLC
Locations (56):
- United States (10):
  - Clinical Research Site 1357, Lincoln, California
  - Clinical Research Site 1358, Long Beach, California
  - Clinical Research Site 1361, San Dimas, California
  - Clinical Research Site 1031, Port Orange, Florida
  - Clinical Research Site 1271, Chicago, Illinois
  - Clinical Research Site 1359, Topeka, Kansas
  - Clinical Research Site 1009, Berlin, New Jersey
  - Clinical Research Site 1037, Trenton, New Jersey
  - Clinical Research Site 1008, Munroe Falls, Ohio
  - Clinical Research Site 1360, San Antonio, Texas
- Czechia (5):
  - Clinical Research Site 3119, Hodonín
  - Clinical Research Site 3123, Mladá Boleslav
  - Clinical Research Site 3120, Olomouc
  - Clinical Research Site 3112, Prague
  - Clinical Research Site 3122, Prostějov
- Hungary (6):
  - Clinical Research Site 9102, Balatonfüred
  - Clinical Research Site 9101, Balatongyörök
  - Clinical Research Site 9106, Budapest
  - Clinical Research Site 9107, Szeged
  - Clinical Research Site 9105, Zalaegerszeg
  - Clinical Research Site 9103, Zamárdi
- Japan (12):
  - Clinical Research Site 6031, Chiba
  - Clinical Research Site 6037, Chiba
  - Clinical Research Site 6042, Chiba
  - Clinical Research Site 6040, Fukuoka
  - Clinical Research Site 6035, Fukuoka
  - Clinical Research Site 6034, Ibaraki
  - Clinical Research Site 6039, Ibaraki
  - Clinical Research Site 6041, Ibaraki
  - Clinical Research Site 6032, Ibaraki
  - Clinical Research Site 6033, Ōsaka
  - Clinical Research Site 6036, Shizuoka
  - Clinical Research Site 6038, Tochigi
- Poland (13):
  - Clinical Research Site 7137, Gdansk
  - Clinical Research Site 7144, Krakow
  - Clinical Research Site 7142, Krakow
  - Clinical Research Site 7139, Krakow
  - Clinical Research Site 7141, Krakow
  - Clinical Research Site 7120, Lublin
  - Clinical Research Site 7138, Lublin
  - Clinical Research Site 7131, Olsztyn
  - Clinical Research Site 7143, Poznan
  - Clinical Research Site 7140, Poznan
  - Clinical Research Site 7136, Poznan
  - Clinical Research Site 7107, Puławy
  - Clinical Research Site 7128, Torun
- Spain (10):
  - Clinical Research Site 9002, Alicante
  - Clinical Research Site 9016, Almería
  - Clinical Research Site 9005, Alzira
  - Clinical Research Site 9017, Barcelona
  - Clinical Research Site 9013, Barcelona
  - Clinical Research Site 9012, Madrid
  - Clinical Research Site 9011, Seville
  - Clinical Research Site 9014, Seville
  - Clinical Research Site 9015, Seville
  - Clinical Research Site 9018, Valencia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Bexagliflozin: Subjects will receive a bexagliflozin tablet, 20 mg, once daily for the duration of the study. Subjects will continue taking metformin and receive placebo for sitagliptin daily for the duration of the study.
  Bexagliflozin: 20 mg, tablet
  Placebo for sitagliptin: 100 mg inactive tablet to match active comparator
- Sitagliptin: Subjects will receive a sitagliptin tablet, 100 mg, once daily for the duration of the study. Subjects will continue taking metformin and receive placebo for bexagliflozin for the duration of the study.
  Sitagliptin: 100 mg, tablet
  Placebo for bexagliflozin: 20 mg inactive tablet to match active comparator
Period: Overall Study
Arm/Group | Bexagliflozin | Sitagliptin
Started | 192 | 194
Intention-to-treat (One randomized subject in each group was excluded in the ITT and the safety populations due to site closure for GCP violation.) | 191 | 193
Completed | 180 | 189
Not Completed | 12 | 5
Not completed — Adverse Event | 5 | 1
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 1 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Site closure | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bexagliflozin | Sitagliptin | Total
Number analyzed (Participants) | 191 | 193 | 384
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (9.69) | 59.6 (9.76) | 59.4 (9.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 67 | 138
  Male | 120 | 126 | 246
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 10
  Not Hispanic or Latino | 188 | 186 | 374
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 27 | 35 | 62
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 2 | 8
  White | 158 | 156 | 314
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Hungary | 33 | 23 | 56
  Czechia | 16 | 25 | 41
  United States | 15 | 21 | 36
  Japan | 27 | 35 | 62
  Poland | 70 | 44 | 114
  Spain | 30 | 45 | 75
Height [Mean (Standard Deviation); unit: cm] | 167.4 (10.67) | 168.3 (9.63) | 167.9 (10.16)
Body Weight [Mean (Standard Deviation); unit: kg] | 90.27 (20.736) | 89.44 (19.235) | 89.85 (19.974)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 32.06 (6.052) | 31.39 (5.294) | 31.72 (5.686)
HbA1c [Mean (Standard Deviation); unit: percentage of glycated hemoglobin] | 7.94 (0.808) | 8.03 (0.921) | 7.99 (0.867)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 24
Description: The primary efficacy objective is to demonstrate that bexagliflozin is non-inferior to sitagliptin by evaluating the treatment effect on hemoglobin A1c (HbA1c) reduction at week 24 in subjects whose type 2 diabetes mellitus (T2DM) is inadequately controlled by metformin.
Time Frame: Baseline to week 24
Population: Subjects in the intention-to-treat population and with a value at baseline and at week 24 were included.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of HbA1c
Arm/Group | Bexagliflozin | Sitagliptin
Number analyzed (Participants) | 180 | 190
percentage of HbA1c | -0.74 [-0.86 to -0.62] | -0.82 [-0.93 to -0.71]
Statistical Analysis 1: Comparison: Bexagliflozin vs Sitagliptin; Test type: Non-Inferiority — The non-inferiority margin of 0.35% was determined based on a reference clinical trial that demonstrated the effectiveness of sitagliptin, 100 mg, compared to placebo on HbA1c reduction in subjects with type 2 DM. A margin of 0.35% was selected to be approximately half of sitagliptin effect and remained clinically meaningful; Difference of LS Means = 0.08, 95% CI 2-sided [-0.07 to 0.22] — Mixed-effects repeated measures analysis includes region, treatment, visit, treatment-by-visit interaction and the baseline HbA1c value as fixed effect covariates

2. Secondary Outcome: Change in FPG From Baseline at Week 24
Description: To evaluate the treatment effect of bexagliflozin vs. sitagliptin on the change in fasting plasma glucose (FPG) at week 24
Time Frame: Baseline to week 24
Population: Subjects in the intention-to-treat population and with values at baseline and at week 24 were included.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Bexagliflozin | Sitagliptin
Number analyzed (Participants) | 180 | 190
mmol/L | -1.82 [-2.09 to -1.55] | -1.45 [-1.70 to -1.19]
Statistical Analysis 1: Comparison: Bexagliflozin vs Sitagliptin; Test type: Superiority; p = 0.0123, Mixed-effects repeated measures; Covariate includes region, treatment, visit, treatment-by-visit interaction and the baseline FPG value as a fixed effect covariate; Difference of LS Means = -0.37, 95% CI 2-sided [-0.70 to -0.05]

3. Secondary Outcome: Change in Body Weight in Subjects With Baseline BMI ≥ 25 kg/m2 at Week 24
Description: To evaluate the treatment effect of bexagliflozin vs. sitagliptin on the change in body weight in subjects with baseline body mass index (BMI) ≥ 25 kg/m2 at week 24
Time Frame: Baseline to week 24
Population: Subjects in the intention-to-treat population with a baseline body mass index >= 25 kg/m2 and had body weight values at baseline and at week 24 were included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Groups:
- Bexagliflozin: Subjects received a bexagliflozin tablet, 20 mg, once daily for the duration of the study. Subjects continued taking metformin and received placebo for sitagliptin daily for the duration of the study.
  Bexagliflozin: 20 mg, tablet
  Placebo for sitagliptin: 100 mg inactive tablet to match active comparator
- Sitagliptin: Subjects received a sitagliptin tablet, 100 mg, once daily for the duration of the study. Subjects continued taking metformin and received placebo for bexagliflozin for the duration of the study.
  Sitagliptin: 100 mg, tablet
  Placebo for bexagliflozin: 20 mg inactive tablet to match active comparator
Arm/Group | Bexagliflozin | Sitagliptin
Number analyzed (Participants) | 158 | 171
kg | -3.35 [-3.85 to -2.84] | -0.81 [-1.29 to -0.32]
Statistical Analysis 1: Comparison: Bexagliflozin vs Sitagliptin; Test type: Superiority; p < 0.0001, Mixed-effects repeated measures; Included region, treatment, visit, treatment-by-visit interaction and the baseline body weight value as fixed effect covariate; Difference of LS Means = -2.54, 95% CI 2-sided [-3.15 to -1.92]

4. Secondary Outcome: Change in SBP in Subjects From Baseline at Week 24
Description: To evaluate the treatment effect of bexagliflozin vs. sitagliptin on the change in systolic blood pressure (SBP) in subjects at week 24
Time Frame: Baseline to week 24
Population: Subjects in the intention-to-treat population with values at baseline and at week 24 were included.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Bexagliflozin | Sitagliptin
Number analyzed (Participants) | 180 | 190
mm Hg | -4.23 [-6.18 to -2.28] | -1.90 [-3.75 to -0.06]
Statistical Analysis 1: Comparison: Bexagliflozin vs Sitagliptin; Test type: Superiority; p = 0.0276, t-test, 1 sided; p value was presented based on one sided statistical tests using a 0.025 level of significance; mixed-effects repeated measures = -2.33, 95% CI 2-sided [-4.70 to 0.05] — Included region, treatment, visit, treatment-by-visit interaction and the baseline body weight value as fixed effect covariate

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from 1 week prior to randomization (V2) until Week 26 (V8/follow up visit)
Arm/Group | Bexagliflozin | Sitagliptin
All-Cause Mortality (participants affected / at risk) | 1/191 | 0/193
Serious Adverse Events (participants affected / at risk) | 7/191 | 4/193
Other Adverse Events (participants affected / at risk) | 28/191 | 47/193
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bexagliflozin (N=191) | Sitagliptin (N=193)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Microvascular coronary artery disease (Cardiac disorders) | 1 (2) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Gallstone ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intracranial aneursym (Nervous system disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bexagliflozin (N=191) | Sitagliptin (N=193)
Nasopharyngitis (Infections and infestations) | 15 (15) | 25 (29)
Influenza (Infections and infestations) | 3 (3) | 10 (10)
Urinary tract infection (Infections and infestations) | 7 (9) | 4 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 6 (12) | 10 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has no right to publish trial results.

DOCUMENTS (2):
  • Study Protocol (2017-04-06): https://cdn.clinicaltrials.gov/large-docs/12/NCT03115112/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/12/NCT03115112/SAP_001.pdf